CLINICAL TRIAL: NCT05501951
Title: Reduce High-risk Behaviours Under Chronic Stress Via tDCS-induced Neural Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LI Cheng (Other)
Responsible Party: Sponsor-Investigator, LI Cheng, Postdoctoral fellow, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCSHKU
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Risk-Taking; Chronic Stress
MeSH Terms: conditions — Risk-Taking | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- right DLPFC tDCS (Experimental): Participants in this group will receive 10 sessions of right DLPFC tDCS
  Interventions: Other: tDCS stimulation
- right OFC tDCS (Experimental): Participants in this group will receive 10 sessions of right OFC tDCS
  Interventions: Other: tDCS stimulation
- Control group (Sham Comparator): Participants in this group will receive 10 sessions of sham stimulation
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: tDCS stimulation — The transcranial direct current stimulation (tDCS) method has emerged in the recent years as a non-invasive, safe, cheap, convenient and effective means to modulate brain functions and behaviours
  Arms: right DLPFC tDCS; right OFC tDCS
Other: Sham stimulation — For the sham group, the electrode positioning will be randomly allocated to be identical to either the DLPFC or the OFC group, and active stimulation will be delivered for the first 30 seconds only
  Arms: Control group

SUMMARY:
The persistent political conflicts and COVID-19 pandemic have led to elevated chronic stress levels in Hong Kong, with far-reaching and profound negative impacts on the citizen's mental health. An important pathway via which chronic stress negatively impacts health is through promoting high-risk behaviours, such as addiction, suicide, and antisocial acts. Therefore, testing means to break the association between chronic stress and high-risk behaviour is essential to reducing the adverse consequences of stress and promoting stress resilience. The transcranial direct current stimulation (tDCS) may be a viable method for reducing risky tendency in high-stress individuals, through modulating brain functions and plasticity. Although single-session tDCS has been shown to reliably reduce risky decision making and behaviours acutely, its efficacy over extended periods of time has not been demonstrated, particularly among non-clinical samples. Being able to show that tDCS could lead to long-lasting reduction of risky tendency is necessary for promoting the wide application of this method in therapeutic settings. In this project, we aim to conduct a randomised control trial to systematically and comprehensively test whether 10 sessions of tDCS on either the dorsolateral prefrontal cortex or the orbitofrontal cortex would lead to reduction in risky tendency not only immediately after treatment, but also at 1 month and 3 months after treatment.

Participants will be healthy male and female adults (21-40 years old) under relatively high levels of chronic stress, as selected from an online survey prior to the study.

Participants will be randomly allocated to one of 3 treatment groups: DLPFC tDCS, OFC tDCS, and sham control. At baseline, participants will complete several risk-taking assessments, including an established computerised task that measures both risk taking and a cognitive bias that was shown to increase irrational risky tendency (illusion of control), an established questionnaire that measures risky decision making in real-life scenarios, and a scale measuring past engagement in common risky activities.

Participants will also complete various personality and mood questionnaires, along with assessments on important cognitive abilities. We hypothesized that both DLPFC and OFC tDCS would reduce risk taking across the 3 timepoints, but the effect of DLPFC tDCS would be mediated by reduction in cognitive bias, whereas that of OFC tDCS would be mediated by increase in inhibition functions. These hypotheses will be tested by linear mixed models and mediation analyses. Additional exploratory analyses also test whether the tDCS effect would be moderated by relevant personality factors such as impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21-40 years;
* Fluent in reading and writing Chinese (Cantonese or Mandarin);
* Right-handed as assessed with the Edinburgh Handedness Inventory;
* Normal or corrected-to-normal vision and hearing;
* IQ>90 as assessed with the Test of Nonverbal Intelligence, 4th edition (TONI-IV)

Exclusion Criteria:

* Past or present physical illness, organic brain disorder, traumatic brain injury, addiction, impulse control disorder, psychotic disorder, affective disorder, or any other major neurological or psychological condition;
* First-degree relative with past or present major psychological disorder or suicidal behaviour;
* Intake of psychotropic medication or any other medication that may affect cognition in the 6 months preceding the study day;
* (For women) being pregnant;
* any contraindication for tDCS, such as having a cerebral implant or history (either personal or family) of seizure. The psychological conditions will be assessed using the Structured Clinical Interview for DSM-5 Disorders-Clinician Version (SCID-5-CV).

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes in risk taking behavior | Baseline; 1-month follow up; 3-month follow up
  Changes in risk taking will be assessed using the IoC card gambling task